CLINICAL TRIAL: NCT06753110
Title: A Multicenter, Multinational, Cohort Long-term Post-market Clinical Follow-up (PMCF) of the Safety and Efficacy of the Osseoanchored Prostheses for the Rehabilitation of Amputees (OPRA) Implant System When Used for Transhumeral Implantation in Amputee Patients
Acronym: ReTHro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0092
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Amputation of Upper Limb
Keywords: Skeletal anchorage of amputation prostheses.; Osseoanchored Prosthesis

STUDY DESIGN:
Intervention Model Description: As described in the title this is a long term safety and efficacy follow up on subjects that received an transhumeral implant uni/bilaterlly before Jan 2024, and mainly looking at Retrospective data gathered from medical records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uni/bilaterally transhumeral amputated (Other): OPRA transhumeral
  Interventions: Device: OPRA transhumeral

INTERVENTIONS:
Device: OPRA transhumeral — Skeletal anchorage of amputation prostheses.

SUMMARY:
This non-interventional clinical investigation is initiated for the purpose of long-term Post-Market Clinical Follow-up (PMCF) and the follow-up time of patients is expected to span from 6 months to >20 years in function. It will collect and evaluate clinical data on the safety and performance of the OPRA™ Implant System when used on transhumeral amputees and within the scope of the intended use.

DETAILED DESCRIPTION:
All subjects that will be enrolled in this investigation should have been treated with the OPRA Implant System for a transhumeral unilateral or bilateral amputation and completed the second stage surgery (S2) and had at least 6 months of usage experience with the OPRA Implant System before enrolment.

This retrospective, non-interventional, clinical investigation is designed as a multicenter, multinational, cohort investigation for long-term follow-up of safety and efficacy endpoints. The investigation will also include prospective visit(s) for enrollment of subjects and collection of present data on device functionality and the use of the device.

No control group or comparator will be used in this investigation.

All patient reported outcome questionnaires used in the investigation will be available at the investigation site for completion by the subjects during one of the subjects' visits to the site. Depending on the subjects' preferences it will also be possible to provide those questionnaires to the subjects, through use of regular mail, email or through an electronic Patient Reported Outcome system (ePRO). It will be possible for the subjects to complete the questionnaires either on paper, electronically or over phone, depending on their preferences.

Preferably, the subjects prosthesis functional tests should be performed as part of the follow-up visit at the site. The tests may also be performed remotely, depending on subjects' preferences. If done remotely, this will require the functionality test being performed during a videoconference with the test administrator. No photos or video-recordings (if conducted according to the sites normal practice) of the performed tests will be part of the investigation documentation, only the related medical record notes will be used as source data for those parameters.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral amputation
* OPRA™ implant system placed, and with S2 completed before 01-Jan-2024
* Having a minimum of 6 months of follow-up between S2 and enrolment

Exclusion Criteria:

* Subject not willing to consent
* Subject implanted with the e-OPRA system at the humeral level.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Implant Safety and Effectivness | 2 years post implant surgery
  Implant safety: * Implant survival rate 2 years post implant surgery. Calculated the number of implants still in situ at time of the follow-up visit, 2 years after completion of implant surgery divided by the number of implants at risk.
  Effectivness: * Change in prosthetic use. Measured as time prosthesis used before implant surgery compared with time prosthesis used at time of the follow-up visit.
  Categorized as:
  * Hours per day
  * Days per week.

SECONDARY OUTCOMES:
Implant Safety | More than 10 years
  • Implant survival rate, after 6 months, and 1-, 5-, 10- and ˃10-years post implant surgery.
  Calculated as the number of implants still in situ after 6 months, 1-, 5-, 10- and ˃10-years after completion of surgery divided by the number of implants at risk
Implant Safety | More than 10 years
  • Implant survival time Measured as the time from completion of surgery to implant loss or time of last observation without known implant loss.
Implant safety | More than 10 years
  • Presence of biological complications
  Measured as the number of the following complications taking place from time of surgery to time of implant loss or time of last observation without known implant loss:
  * Infections
  * Skin complications
  * Skeletal complications
Implant safety | More than 10 years
  • Presence of Mechanical complications
  Mechanical complications related to implant, abutment or abutment screw. Measured as the number of mechanical complications taking place from time of surgery to implant loss our time of last observation without known implant loss, presented per category:
  * Implant related
  * Abutment related
  * Abutment screw related
Implant effectiveness | 6 months, 1yr, 2yrs, 5yrs, 10yrs, > 10yrs
  • Functionality evaluations. Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) Set of questions, score 1-5. Higher score worse.
Implant effectiveness | 6 months, 1yr, 2yrs, 5yrs, 10yrs, >10yrs
  Funtionallity evaluation. Patient-Reported Outcomes Measurements Information System(PROMIS) - Upper Extremity, Short Form 7a.
  Seven questions, score 5-1. Higher score better.
Implant effectivness | 6 months, 1yr, 2yrs, 5yrs, 10yrs, >10yrs
  Functionality evaluation. Southampton Hand Assessment Procedure (SHAP). Funtionality test performed, time meassured. Calculated score 0-100. Higher score better.
Implant effectiveness | Through study completion, an avarage of approximately 1 month.
  • Physical evaluation - Short Form (36) Health Survey Eleven questions. Various alternatives.
Implant effectivness | Through study completion, an avarage of approximately 1 month.
  Physical evaluation. Range of Motion Test. Degree of movement around a joint. Higher score better
Implant effectivness. | Through study completion, an avarage of approximately 1 month.
  Physical examination. Pain questions. Numeric Range Scale 0-10. High scores mean worse.
Implant effectiveness | Through study completion, an avarage of approximately 1 month.
  • Satisfaction of use. Prosthetic use satisfaction. Numeric rating scale, 0-10. High score are better.
Implant effectivness | Through study completion, an avarage of approximately 1 month.
  Satisfaction of use. OPRA™ implant system satisfaction. Numeric rating scale, 0-10. High score are better.
Implant effectiveness | Through study completion, an avarage of approximately 1 month.
  • Level of embodiment of the Prosthesis Numerical Rating Scale. Six personal questions. Score 0-10. Second question is 0 better. For the five other question 10 is better.

CONTACTS AND LOCATIONS:
Locations (6):
- The Alfred Hospital, Melbourne, Victoria, Australia
- Medical University of Vienna Clinical laboratory for bionic limb reconstruction Währinger Gürtel 18-20 1090 Vienna, AUSTRIA, Vienna, Austria
- University Hospital Ghent, UX Ghent, Ghent, Belgium
- Germany (2):
  - Hannover Medical School, Hanover
  - University Hospital Tübing, Tübingen
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data specified in the outcome meassures
Supporting Information: SAP, CSR
Time Frame: 2026
Access Criteria: The participating investigators will have full access of the Clinical Investigation Report as part of the study file for archiving. After main publication is performed, individual investigators will have access to the complete data on request.